CLINICAL TRIAL: NCT07268092
Title: Impact of Porcine Extracellular Matrix Nerve Wrap on Spinal Accessory Nerve in Patients Undergoing Neck Dissection for Head and Neck Cancer
Brief Title: Porcine Extracellular Matrix Nerve Wrap in Neck Dissection for Head and Neck Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr Tam have collected the first 20 patients for interim analysis per the protocol, and are trying to get these data to perform interim analyses on these data to best understand how to move forwards.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Samantha Tam, Vice Chair-Otolaryngology • Otolaryngology, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HFHS-1901
Record Dates: First submitted 2025-07-09; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Neck Dissection; Postoperative Complications
Keywords: Spinal Accessory Nerve Injury; Shoulder Dysfunction; Head and Neck Cancer; Nerve Compression Syndromes; Postoperative Complications
MeSH Terms: conditions — Head and Neck Neoplasms; Postoperative Complications; Accessory Nerve Injuries; Nerve Compression Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Arm - Neck dissection with AxoGuard Nerve Protector™ (Experimental): Participants undergo neck dissection surgery for head and neck cancer, during which the spinal accessory nerve (SAN) is wrapped with the AxoGuard Nerve Protector™ (porcine extracellular matrix nerve wrap). This intervention aims to improve postoperative shoulder function by protecting and supporting the nerve during healing. Postoperative physical therapy evaluations will be conducted at baseline, immediate post-op, 1, 6, and 12 months.
  Interventions: Device: Porcine Extracellular Matrix Nerve Wrap (AxoGuard Nerve Protector™)
- Control Arm - Neck dissection without AxoGuard Nerve Protector™. (No Intervention): Participants undergo standard neck dissection surgery for head and neck cancer without the application of the AxoGuard Nerve Protector™. Postoperative physical therapy evaluations will be conducted at baseline, immediate post-op, 1, 6, and 12 months to assess shoulder function.

INTERVENTIONS:
Device: Porcine Extracellular Matrix Nerve Wrap (AxoGuard Nerve Protector™) — The intervention involves the application of the AxoGuard Nerve Protector™, a nerve wrap derived from porcine extracellular matrix (ECM), to the spinal accessory nerve (SAN) during neck dissection surgery in head and neck cancer patients. The device is designed to protect and support the nerve by preserving the extracellular matrix and creating a favorable environment for nerve healing. This helps prevent inflammation and fibrosis around the nerve, potentially improving postoperative shoulder function. The nerve wrap is applied intraoperatively after dissection but before surgical closure. The study compares this intervention to standard neck dissection without nerve wrapping.
  Arms: Treatment Arm - Neck dissection with AxoGuard Nerve Protector™

SUMMARY:
Perform a preliminary efficacy study using the porcine extracellular matrix nerve wrap (AxoGuard Nerve Protector™, AxoGen Inc., Alachua, FL) to wrap the spinal accessory nerve (SAN) during neck dissections for head and neck cancer as it relates to postoperative shoulder function, both subjectively and objectively.

DETAILED DESCRIPTION:
Many patients who have surgery for head and neck cancer also need a procedure called a neck dissection, where lymph nodes and tissue are removed from the neck. During this surgery, even when a nerve called the spinal accessory nerve (SAN) is carefully preserved, patients often have shoulder problems afterward. These problems can include pain, weakness, and difficulty lifting the arm, which can affect daily activities and quality of life.

This study is testing whether using a special nerve wrap made from pig tissue (called AxoGuard® Nerve Protector) can help protect the spinal accessory nerve during surgery and improve shoulder movement and strength after surgery. This nerve wrap is already used in other types of nerve surgeries and may help the nerve heal better by reducing scar tissue and irritation.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients with no previous treatment of head and neck cancer
* Patients with no prior neck surgeries
* Patients undergoing level IIA and IIB neck diss

Exclusion Criteria:

* Patients with previously treated head and neck cancers
* Patients undergoing level V neck dissection
* Patients undergoing bilateral neck dissection
* Patients with previous neck surgery unrelated to head and neck cancer
* Patients allergic to porcine products or with religious/cultural restrictions on porcine products
* Patients unable to consent
* Individuals who are not adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in shoulder flexion active range of motion (degrees) | From preoperative baseline assessment up to 12 months post-surgery
  Shoulder flexion active range of motion will be measured using goniometry. A clinically significant decline is defined as a ≥12° decrease compared to preoperative baseline.
  Unit of Measure: Degrees
Change from baseline in Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) score | From preoperative baseline assessment up to 12 months post-surgery
  Subjective upper extremity function will be assessed using the QuickDASH questionnaire (0-100 scale, higher scores indicate worse disability).
  Unit of Measure: Score
Change from baseline in Neck Dissection Impairment Index (NDII) score | From preoperative baseline assessment up to 12 months post-surgery
  Subjective shoulder-related quality of life will be assessed using the NDII questionnaire (0-50 scale, higher scores indicate greater impairment).
  Unit of Measure: Score
Change from baseline in shoulder abduction active range of motion (degrees | From preoperative baseline assessment up to 12 months post-surgery
  Shoulder abduction active range of motion will be measured using goniometry. A clinically significant decline is defined as a ≥23° decrease compared to preoperative baseline.
  Unit of Measure: Degrees

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Tam, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No